CLINICAL TRIAL: NCT01906229
Title: Acute Pulmonary and Systemic Inflammation in Mechanically Ventilated Intensive Care Patients
Brief Title: Lung and Systemic Inflammation in the Critically Ill Patient
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment and therefore not possible to reach the estimated enrollment
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ronni R. Plovsing, MD, Rigshospitalet, Denmark
Other Study IDs: 959521891
Record Dates: First submitted 2013-07-16; First posted 2013-07-24 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Systemic Inflammatory Response Syndrome (SIRS); Sepsis
MeSH Terms: conditions — Respiratory Distress Syndrome; Systemic Inflammatory Response Syndrome; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Acute respiratory distress syndrome (ARDS)
- Systemic inflammatory response syndrome (SIRS)
- ARDS+SIRS

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a devastating form of acute lung inflammation, that may be caused by a variety of insults with pulmonary and systemic infectious disease being the most common predisposing factor. Sepsis, on the other hand, represents the systemic inflammatory response to an invading pathogen, which may inflict damage upon the host through organ dysfunction. ARDS and sepsis are heterogenous clinical conditions that have a high mortality, and both diseases involve a complex interplay of different inflammatory mediators and cell types. It has been suggested that locally released inflammatory mediators pass from the lungs into the bloodstream following ARDS, triggering systemic inflammation. Conversely, it is possible that severe systemic inflammation may lead to ARDS by an influx of inflammatory mediators from the bloodstream to the lungs. However, the time course and the possible pathways for this transmission of disease have yet to be established.

Investigators hypothesize that:

1. Primary systemic inflammation is followed by a secondary pulmonary inflammatory response
2. Primary pulmonary inflammation is followed by a secondary systemic inflammatory response
3. Both primary and secondary inflammatory responses are characterized by the appearance of pro-inflammatory cytokines, inflammatory cells and production of collagen-like proteins (termed 'lectins')
4. The inflammatory response is most pronounced in the primary afflicted compartment.

ELIGIBILITY:
Inclusion Criteria:

General:

* Age >18 years
* Mechanically ventilated
* < 48 hours after admission to the Intensive Care Unit

Specific:

-ARDS: acute (< 1 week) respiratory failure, characterized by hypoxemia (PaO2/FiO2 < 300 mmHg/40kPa), and bilateral infiltrates on x-ray or CT of thorax, that can not be explained by heart failure og overhydration.

OR

- SIRS (two of the following): Temperature > 38°C or < 36°C, heart rate > 90/min, respiratory frequency > 20 or PaCO2 < 4.2 kPa, leukocytosis (> 12x10^9/L) or leukopenia (< 4x10^9/L)

OR

ARDS + SIRS

Exclusion Criteria:

One lung ventilation; Tube size < 8.0 mm; INR > 1.5 or thrombocytes < 40x10^9/L; Intracranial hypertension; Malignant arrythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Tumor necrosis factor alpha (TNF-a) bioactivity | Day one
Tumor necrosis factor alpha (TNF-a) bioactivity | Day three
Tumor necrosis factor alpha (TNF-a) bioactivity | Day seven
Tumor necrosis factor alpha (TNF-a) bioactivity | Day fourteen

SECONDARY OUTCOMES:
Interleukin (IL)-6 | Day one
Mannose binding lectin (MBL) | Day one
Ficolin-1,2,3 | Day one

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit, 4131, Rigshospitalet, Copenhagen Ø, Denmark